CLINICAL TRIAL: NCT01749436
Title: Role of Lung Ultrasound Imaging for Intraoperative Monitoring of Atelectasis During Laparoscopic Surgery
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Other Study IDs: MG2012-001
Record Dates: First submitted 2012-12-12; First posted 2012-12-13 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Atelectasis
Keywords: Atelectasis; Pneumoperitoneum; Hypoxemia
MeSH Terms: conditions — Pulmonary Atelectasis; Pneumoperitoneum; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lung ultrasound imaging: Lung ultrasound imaging examinations performed during the perioperative period for the monitoring of atelectasis associated with laparoscopic surgery
  Interventions: Other: Lung ultrasound imaging examinations

INTERVENTIONS:
Other: Lung ultrasound imaging examinations — Lung ultrasound examinations performed at different time-points immediately before surgery, during surgery under general anesthesia and after surgery in the recovery room to detect and monitor atelectasis related to laparoscopic procedures.

SUMMARY:
General anesthesia results in the development of atelectasis in the dependent areas of the lungs exposing patients to an increased risk of hypoxemia. During laparoscopic procedures, pneumoperitoneum increases already present atelectasis.

Several methods have been suggested to reduce the impact of atelectasis during surgery. However, few intraoperative modalities for the diagnosis and monitoring of atelectasis are available. Lung ultrasound imaging is a promising non-invasive, non-radiant, portable and easy to use tool that as yet to be studied in the intraoperative setting.

This observational study will aim to clarify the role of lung ultrasound imaging during laparoscopic surgery for the diagnostic and monitoring of atelectasis.

This study is designed to:

* Demonstrate a link between the lung ultrasound aeration score, the partial pressure of oxygen in arterial blood (PaO2) / fraction of inspired oxygen (FiO2) ratio and the oxygenation index.
* In the event of intraoperative desaturation, study the impact of positive end-expiratory pressure (PEEP) and/or increase of FiO2 on the aeration score.
* Study the impact of pain on diaphragmatic function and the aeration score.

Our hypothesis is that lung ultrasound imaging allows detection of lung aeration changes associated with induction of general anesthesia, pneumoperitoneum, emergence from anesthesia and changes occurring during the stay in the recovery room.

DETAILED DESCRIPTION:
On arrival in the operating theatre, each patient will undergo a baseline lung ultrasound examination.

The anesthetic technique and monitoring will be standardized. The radial artery will be cannulated after induction of anesthesia for blood gas monitoring.

Lung ultrasound examinations will be performed 5 minutes following induction of general anesthesia and 5 minutes after insufflation of the abdomen with carbon dioxide. In the event of a desaturation needing an intervention (increase of FiO2 or PEEP), ultrasound imaging will be repeated before and after the intervention. Presence of a pneumothorax or endobronchial intubation will be assessed during each examination. Fifteen minutes after arrival and immediately before discharge from the recovery room, lung ultrasound examinations will also be performed.

FiO2 and vital signs will be recorded at each ultrasound examination. Arterial blood samples will be collected simultaneously. Pain rating using the visual analog scale and diaphragmatic function will be assessed during the preoperative ultrasound examination and before discharge from the recovery room.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Scheduled for laparoscopic surgery
* Physical status 1-3

Exclusion Criteria:

* Previous thoracic procedure (thoracic drain, thoracotomy, thoracoscopy)
* Contraindication to the placement of an arterial line
* Very severe chronic obstructive pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for laparoscopic surgery
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Lung aeration | From arrival in the operating theatre to immediately before discharge from the recovery room (Day 0)
  Estimate lung aeration by ultrasound imaging using a four point aeration score (0 = normal lung, 1 = moderate aeration loss, 2 = severe aeration loss, 3 = complete aeration loss and consolidation)

SECONDARY OUTCOMES:
Gas exchange | From 5 minutes following induction of anesthesia to immediately before discharge from the recovery room (Day 0)
  Assess the impact of the different stages of anesthesia and surgery on gas exchange by measuring arterial blood gases.
Diaphragmatic function | On arrival in the operating theatre and immediately before discharge from the recovery room (Day 0)
  Assess diaphragmatic function by ultrasound imaging
Incidence of pneumothorax | From 5 minutes following induction of anesthesia to immediately before discharge from the recovery room (Day 0)
  Estimate the incidence of pneumothorax by ultrasound imaging
Incidence of endobronchial intubation | From 5 minutes following induction of anesthesia to immediately before discharge from the recovery room (Day 0)
  Estimate the incidence endobronchial intubation by ultrasound imaging

CONTACTS AND LOCATIONS:
Overall Officials: Martin Girard, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada